CLINICAL TRIAL: NCT00174772
Title: A Two Arm Phase II Study Comparing Docetaxel/Cisplatin Induction Therapy Followed By Concurrent Chemoradiotherapy Versus Concurrent Chemoradiotherapy Followed By Consolidation Docetaxel/Cisplatin in Patients With Locally Advanced Unresectable NSCLC (Stage IIIA-Multiple cN2 or IIIB)
Brief Title: Pulmonart: Docetaxel - Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_2505
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Cisplatin; Radiotherapy

ARMS (2):
- B (Experimental): Concurrent chemoradiotherapy followed by consolidation chemotherapy
  Interventions: Drug: docetaxel and cisplatin + radiotherapy followed by docetaxel and cisplatin
- A (Experimental): Induction chemotherapy followed by concurrent chemoradiotherapy
  Interventions: Drug: docetaxel and cisplatin followed by concurrent chemoradiotherapy with docetaxel and cisplatin + radiotherapy

INTERVENTIONS:
Drug: docetaxel and cisplatin followed by concurrent chemoradiotherapy with docetaxel and cisplatin + radiotherapy — docetaxel (75mg/m2, IV, Day 1) and cisplatin (40 mg/m2, IV, Day 1, 2) every 3 weeks for 2 cycles, followed by concurrent chemoradiotherapy with docetaxel (20 mg/m2, IV) and cisplatin (20 mg/m2) weekly for 6 weeks + radiotherapy 2 Gy/day, 5 days per week to a total dose of 66 Gy
  Arms: A
Drug: docetaxel and cisplatin + radiotherapy followed by docetaxel and cisplatin — docetaxel (20mg/m2, IV) and cisplatin (20 mg/m2) weekly for 6 weeks + radiotherapy 2 Gy/day, 5 days per week to a total dose of 66 Gy followed by docetaxel and cisplatin (40 mg/m2, IV, Day 1, 2) every 3 weeks for 2 cycles.
  Arms: B

SUMMARY:
Primary Objective:

* To evaluate the toxicity/safety profile of docetaxel/cisplatin induction therapy followed by concurrent chemoradiotherapy versus concurrent chemoradiotherapy followed by consolidation docetaxel/cisplatin in patients with locally advanced unresectable NSCLC (stage IIIA- multiple cN2 or IIIB).

Secondary Objective:

* To estimate efficacy parameters in overall response rate, progression free survival and 1 year survival for each of the two above mentioned arms.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma or a combination of these)
* Patients must have a locoregionally advanced unresectable NSCLC

  * Stage IIIA with multiple level clinical N2 nodes (preferably with histological or cytological confirmation).
  * Patients with peripheral tumours of the lower lobe with contralateral upper mediastinal nodes at station N2 are excluded
  * Stage IIIB T4 or N3

    * In the T4 category, patients with pleural or pericardial effusion and multiple nodules in the same lobe are excluded.
    * Patients with T4 disease secondary to extensive and massive involvement of the great vessels are excluded.

Patients should be excluded when the expected risk of pulmonary toxicity is likely to be high, e.g. V20 in excess of 35%.

* Life expectancy of at least 12 weeks.
* WHO performance status 0 or 1.
* Weight loss ≤ 10% within the last 3 months.
* Laboratory requirements at entry (within 7 days before randomization):

  * Blood cell counts:

    * Absolute neutrophils ≥ 2.0 x 10^9/L
    * Platelets ≥ 100 x 10^9/L
    * Hemoglobin ≥ 10 g/dl
  * Renal function:

    _Serum creatinine ≤1 x the upper limit of normal (UNL). In case of borderline value of serum creatinine, the 24h creatinine clearance should be ≥ 60 mL/min
  * Hepatic functions:

    * Serum bilirubin ≤ 1 x UNL
    * ASAT and ALAT ≤ 2.5 x UNL
    * Alkaline phosphatase ≤ 5 x UNL.

Patients with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.

* Lung function tests at entry:

  * FEV1: ≥ 50 % x Normal value
  * DLco: ≥ 50 % x Normal value.
* Adequate cardiac function.
* Patient with either measurable and/or non-measurable lesion (according to RECIST criteria).

Exclusion criteria:

* Diagnosis of small cell lung cancer
* Pregnant or lactating women
* Patients (male or female) with reproductive potential not implementing adequate contraceptive measures
* Prior systemic chemotherapy, immunotherapy, or biological therapy including neoadjuvant or adjuvant treatment for NSCLC
* Prior surgery for NSCLC, if less than 5 years from study
* Prior radiotherapy for NSCLC
* History of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years.
* Symptomatic peripheral neuropathy Grade ≥ 2 except if due to trauma.
* Other serious concomitant illness of medical conditions:

  * Congestive heart failure or angina pectoris except if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmias.
  * History of significant neurologic or psychiatric disorders including dementia or seizures.
  * Active infection requiring IV antibiotics.
  * Active ulcer, unstable diabetes mellitus or other contra-indication to corticosteroid therapy.
  * Superior vena cava syndrome contra-indicating hydration.
  * Preexisting pericardial effusion.
  * Preexisting symptomatic pleural effusion.
* Significant gastrointestinal abnormalities, including requirement for intravenous nutrition, active peptic ulcer disease, prior surgical procedures affecting absorption.
* Distant metastasis.
* Concurrent treatment with any other experimental anti-cancer drugs.
* Concomitant or within 4-week period administration of any other experimental drug under investigation.
* Significant ophthalmologic abnormalities.
* Moderate to severe dermatitis.
* Hypersensitivity to docetaxel or any of its excipients.
* Concomitant use of phenytoin, carbamazepin, barbiturates, or rifampicin.
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Patient unlikely to comply with protocol, i.e., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
anti-tumor activity including overall response rate | assessed at the end of the full course of treatment period

SECONDARY OUTCOMES:
all treatment related acute and chronic toxicity assessed according to the NCI-CTC scale | throughout the study
other adverse events not reported in the NCI-CTI scale | throughout the study
hematological and non-hematological toxicities | reported for all grades observed during each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Background] van Sornsen de Koste JR, Senan S, Underberg RW, Oei SS, Elshove D, Slotman BJ, Lagerwaard FJ. Use of CD-ROM-based tool for analyzing contouring variations in involved-field radiotherapy for Stage III NSCLC. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):334-9. doi: 10.1016/j.ijrobp.2005.02.016. PMID 16168828